CLINICAL TRIAL: NCT01249599
Title: Stress-induced Vascular Dysfunction: Evaluation of Endothelial Function in a Cohort of Patients With Takotsubo Syndrome
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0210/1
Record Dates: First submitted 2010-11-22; First posted 2010-11-30 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Takotsubo Syndrome
Keywords: Takotsubo Syndrome; apical balooning syndrome; stress-cardiomyopathy; endothelial function; sympathetic nervous activity; platelet adhesion; arterial compliance
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: blood sample analysis — The aim of this prospective single-center study is to evaluate endothelial function, vascular compliance, oxidative stress parameters, quality of life and platelet adhesion in patients with apical ballooning syndrome and age-matched controls.

SUMMARY:
The aim of this prospective single-center study is to evaluate endothelial function, arterial compliance, sympathetic nervous activity at rest and after mental and physical stress, carotid atherosclerosis, oxidative stress parameters, quality of life and platelet adhesion in patients with apical ballooning syndrome and age-matched controls.

DETAILED DESCRIPTION:
The aim of this prospective single-center study is to evaluate endothelial function, arterial compliance, sympathetic nervous activity at rest and after mental and physical stress, carotid atherosclerosis, oxidative stress parameters, quality of life and platelet adhesion in patients with Takotsubo Syndrome (apical ballooning syndrome/broken heart syndrome) and age-matched controls.

ELIGIBILITY:
Inclusion criteria: We plan to include male or female subjects, age 18-80 with a diagnosis of Takotsubo Syndrome (according to standard clinical criteria[Strony, J., et al., Analysis of shear stress and hemodynamic factors in a model of coronary artery stenosis and thrombosis. Am J Physiol, 1993. 265(5 Pt 2): p. H1787-96.]) in the last 10 years.

Moreover, patients matched to the Takotsubo patients for age and cardiovascular risk factors will be included in the control group.

All patients will signed an written informed consent

Exclusion criteria:

* Long acting nitrates, or PDE-5-Hemmer
* Alcohol or drug abuse,
* Malignancy (unless healed or remission > 5 years)
* Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
* Pulmonary Hypertension
* Participation in another study within the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female subjects, age 18-80 with a diagnosis of Takotsubo Syndrome according to standard clinical criteria [Strony, J., et al., Analysis of shear stress and hemodynamic factors in a model of coronary artery stenosis and thrombosis. Am J Physiol, 1993. 265 (5 Pt 2): p. H1787-96.] in the last 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Endothelial function as flow mediated dilatation | baseline
  Evaluation of endothelial function as flow mediated dilation in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors

SECONDARY OUTCOMES:
Evaluation of vascular compliance as pulse wave analysis | baseline
  Comparison of vascular compliance as pulse wave analysis in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Evaluation of pulse wave velocity | baseline
  Comparison of pulse wave velocity in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Evaluation of carotid atherosclerosis as intima-media-thickness and total plaque area | baseline
  Comparison of carotid atherosclerosis as intima-media-thickness and total plaque area in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Measurement of sympathetic nervous activity | baseline
  Comparison of sympathetic nervous activity at rest, after cold pressor test and after mental stress tests in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Evaluation of platelet adhesion | baseline
  Comparison of shear-stress dependent platelet adhesion by the Cone and Platelet Analyzer in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Evaluation of oxidative stress parameters | baseline
  Comparison of oxidative stress parameters in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Evaluation of tissue factor plasma level | baseline
  Comparison of tissue factor plasma level in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors
Assessment of quality of life and perceived stress, anxiety and depression | baseline
  Comparison of "quality of life" and "perceived stress, anxiety and depression" in patients with apical ballooning syndrome and controls matched for age and cardiovascular risk factors Quality of life will be assessed using the German version of the European Quality of Life Questionnaire EQ-5D (www.euroqol.org). Perceived stress, anxiety and depression will be assessed by the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Noll, Prof MD, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Naegele M, Flammer AJ, Enseleit F, Roas S, Frank M, Hirt A, Kaiser P, Cantatore S, Templin C, Frohlich G, Romanens M, Luscher TF, Ruschitzka F, Noll G, Sudano I. Endothelial function and sympathetic nervous system activity in patients with Takotsubo syndrome. Int J Cardiol. 2016 Dec 1;224:226-230. doi: 10.1016/j.ijcard.2016.09.008. Epub 2016 Sep 12. PMID 27661411